CLINICAL TRIAL: NCT02645162
Title: A Cluster Randomized Control Trial to Evaluate the Efficacy and Feasibility of a Community-based Preschool Programme and Community Engagement Strategy Led by Community Youth Leaders in Rural Pakistan
Brief Title: Youth Leaders for Early Childhood Assuring Children Are Prepared for School
Acronym: LEAPS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Grand Challenges Canada (Other); UNICEF (Other); Yale University (Other)
Responsible Party: Principal Investigator, Dr Aisha Khizar Yousafzai, Dr., Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3450-PED-ERC-15
Record Dates: First submitted 2015-12-31; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Child Development
Keywords: Pakistan; Early Child Development, Care and Education; Youth Leaders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preschool (Experimental): * This arm will receive the community-based preschool intervention.
  * The preschool sessions will include 2 groups per day (3 years 6months to 4 years 6 months in the morning session and 4 years 7 months to 5 year 6 months in the afternoon session at the time of enrolment)
  * Each session will last 3 hours for 5 days per week.
  * The expected CYL-to-child ratio will be 1:15; however, given the expected high level of local demand it may exceed to a maximum of 1:20 ratio.
  Interventions: Behavioral: Community-based Preschool
- Control (No Intervention): The control group will receive standard services available in the community.

INTERVENTIONS:
Behavioral: Community-based Preschool — * Preschool sessions in community-based preschool
  * Run by trained community youth leaders from the same village.
  Arms: Preschool

SUMMARY:
Worldwide about 88 million children drop out of primary school annually. One of the contributory factors is a lack of school readiness among young children, their families and their teachers. To better prepare young children for school, investment in early childhood interventions is necessary. Young children require good health, adequate nutrition and social-emotional, cognitive and communication skills to succeed in school, which requires both support in the family environment and a stable transition to the classroom environment. Preschool programmes are designed to prepare children for formal learning. However, in many low- and middle-income countries there is poor access to quality preschool programmes. Further, the scale-up of early childhood interventions is challenged by a number of barriers such as poor supply (e.g. policy provisions, financing, distance, early child development workforce), inadequate cross-sector coordination, low demand (e.g. knowledge mobilization, agency, community of purpose, opportunities to participate) and weak quality of services (e.g. training, supervision and monitoring systems).

In partnership with the National Commission for Human Development, we propose to implement an early childhood care and education programme in rural Sindh that is championed by Community Youth Leaders. The Community Youth Leaders will run community preschools for children aged 3-6 years, and will also coordinate local community engagement and local stakeholder strategies across sectors to leverage demand-side actions to promote ownership and scale-up of early childhood interventions. The LEAPS Programme (Youth Leaders for Early Childhood Assuring Children are Prepared for School) will be evaluated by a cluster randomized controlled efficacy trial. The primary outcome will be children's school readiness, indexed by both early academic and social emotional competencies assessed following 6-9 months of intervention exposure. The compliance, fidelity and quality of the implementation process will also be assessed in order to understand how these features moderate outcomes and whether community-engagement strategies facilitate demand-side actions for scale-up. The expected outcomes for this trial will include a model for quality preprimary education that addresses a current supply-side gap, and will facilitate learning for demand-side actions to support scale-up across a broad range of early childhood interventions.

DETAILED DESCRIPTION:
Trial Design The study is a cluster randomized controlled trial.

Aims Aim 1: To evaluate the effectiveness of the LEAPS Programme on school readiness of children, CYLs, families and services 1.1: To determine whether children who participate in LEAPS preschools led by CYLs will achieve significantly better scores in assessments of school readiness indexed by motor development, social-emotional development, emergent literacy and language, emergent numeracy, approaches to learning and executive functions than children in a control group.

1.2: To identify the moderating and mediating variables (child, CYL, family and community characteristics) for school readiness outcomes among children enrolled in LEAPS preschools.

1.3: To describe the effects of intervention on CYLs' knowledge (ECD and education), competencies (approaches to teaching) and personal/professional growth (executive functioning, aspirations for parenting, family life and career, and autonomy).

1.4: To determine whether LEAPS community engagement strategies to address barriers to scale-up of ECD programmes are effective with respect to family engagement with preschool, support and intent for timely primary school enrolment, family utilization of child services, service provider coordination, knowledge, participation in demand-side platforms and demand-side creation.

Aim 2: To evaluate fidelity and compliance to the LEAPS Programme among community stakeholders 2.1: To evaluate the fidelity of implementation and compliance to the LEAPS preschool programme by the participants.

2.2: To explore stakeholder experience of the preschool programme and community-based strategies to understand facilitators, challenges and learn lessons for scale.

Aim 3: To determine the cost effectiveness of the LEAPS Community-based preschool and community engagement strategies on children's and community readiness for learning and school.

Clusters Ten clusters were randomly selected from a list of 20 clusters part of Responsive Stimulation arm (Yousafzai, A. K., Rasheed, M. A., Rizvi, A., Armstrong, R., & Bhutta, Z. A.. Effect of integrated responsive stimulation and nutrition interventions in the Lady Health Worker programme in Pakistan on child development, growth, and health outcomes: a cluster-randomised factorial effectiveness trial. The Lancet, 384(9950), 1282-1293. 2014) using A-cluster software. Strata were rural/peri-urban. The inclusion criteria of including the cluster in the randomization were: a functioning LHW and a functioning primary school in the village. Five clusters were assigned each for intervention and control arms via simple randomization.

Sample Size The sample size has been estimated as 30 children per cluster with a total of 300 children, which will be adequate taking into account an estimated 10% attrition rate.

Subject Enrolment Control Arm: Children of age as defined by inclusion criteria will be identified from a list of registered children with the Lady Health Worker (nearest record possible). The sample will be stratified by the same age groups as described for the intervention group.

Experimental Arm: A list of children meeting the inclusion criteria was available from the LHW. Any additional child will be verified with the respective LHW prior to enrolment. Enrolment for children in experimental group is defined as child having registered and attended at least 3 days of preschool in week 1.

Data Collection Instruments All instruments were developed in English in the first instance and then translated to Sindhi (with back translations) and piloted prior to use in the study. A systematic adaptation protocol was followed.

Quality Assurance The following strategies are being used

* A 10% sample of assessments are being observed by the field supervisor and scored simultaneously for inter-rater agreement. This shall be followed by a feedback session with the assessor.
* Daily debriefing meetings are held where challenges and solutions will be discussed and will also be used as an opportunity for learning.
* A 10% sample of classroom observations are being video recorded for coding by experts.
* Anthropometry equipment is calibrated daily.

Data Management Forms are being checked prior to entry. The data entry softwares include checks to minimize errors. Data entry is being done at the data entry office located at the field office. All forms are being data entered. A weekly report on status of data entry is being shared by the data entry office.

Data Analysis Plan: An intention to treat model.

ELIGIBILITY:
Inclusion Criteria:

* Resident of study cluster
* Not enrolled in a preschool

Exclusion Criteria:

* Obvious disability

Ages: 42 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
School readiness as defined by the percentage of items passed on a measure of school readiness. | After a minimum of 6 months of intervention exposure.
  Cognitive, social-emotional, motor, early literacy and early numeracy
Child executive functioning tasks composite score | After a minimum of 6 months of intervention exposure
  Inhibitory control, cognitive flexibility, working memory

OTHER OUTCOMES:
Knowledge and Practice for Health, Hygiene and Nutrition | After a minimum of 6 months of intervention exposure
  Child Report Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aisha K Yousafzai, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yousafzai AK, Rasheed MA, Rizvi A, Shaheen F, Ponguta LA, Reyes CR. Effectiveness of a youth-led early childhood care and education programme in rural Pakistan: A cluster-randomised controlled trial. PLoS One. 2018 Dec 19;13(12):e0208335. doi: 10.1371/journal.pone.0208335. eCollection 2018. PMID 30566498